CLINICAL TRIAL: NCT02055417
Title: Increasing Motivation for Antiretroviral Therapy Initiation: A Pilot Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Melanie Bennett, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00047473
Record Dates: First submitted 2014-02-02; First posted 2014-02-05 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: HIV
MeSH Terms: interventions — Seroconversion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personal Approaches to Treatment Choices for HIV (Experimental): PATCH is a brief intervention designed to support participants' decision-making processes and enhance intrinsic motivation to initiate ART.
  Interventions: Behavioral: Personal Approaches to Treatment Choices for HIV
- Stress Reduction Skills Program (Active Comparator): SRSP includes training in stress reduction skills such as relaxation, problem solving, and expressing negative feelings.
  Interventions: Behavioral: Stress Reduction Skills Program

INTERVENTIONS:
Behavioral: Personal Approaches to Treatment Choices for HIV
  Other Names: PATCH
  Arms: Personal Approaches to Treatment Choices for HIV
Behavioral: Stress Reduction Skills Program
  Other Names: SRSP
  Arms: Stress Reduction Skills Program

SUMMARY:
In this 3-year study, the investigators will develop and pilot test an intervention called Personal Approaches to Treatment Choices for HIV (PATCH). PATCH is a brief intervention designed to support participants' decision-making processes and enhance intrinsic motivation to initiate ART, using motivational interviewing (MI) techniques. The intervention will be targeted at HIV-positive African-American adults in inner-city Baltimore, Maryland who are suboptimally engaged in care and who endorse conspiracy beliefs about HIV or low readiness to begin ART. The specific aims are: (1) Develop and refine a manual for a brief MI intervention to support ART decision-making and reduce the likelihood of ART refusal: (2) Evaluate the feasibility and acceptability of implementing the PATCH intervention in a small sample of individuals who are African-American, recommended for ART but who are not current taking it, and who experience multiple barriers to ART adherence; and (3) Conduct a small randomized controlled pilot to test the potential efficacy of the PATCH intervention in producing positive attitudinal changes, including a reduction in conspiracy beliefs and perceived barriers to ART and stated readiness to begin ART.

DETAILED DESCRIPTION:
Many persons with HIV refuse recommended treatment or delay initiation of antiretroviral therapy (ART). Widespread belief in conspiracy theories regarding the origin and treatment of HIV may complicate the ART decision-making process. Research has found that conspiracy beliefs and mistrust in the mainstream medical system are common among African-Americans attending an HIV primary care clinic and that conspiracy beliefs are more likely to be held by patients who are not on ART. Moreover, research shows that conspiracy beliefs and other maladaptive cognitions predict subsequent readiness to begin ART. The investigators have developed an intervention called PATCH: Personal Approaches to Treatment Choices for HIV. PATCH is a brief intervention designed to support participants' decision-making processes and enhance intrinsic motivation to initiate ART, using motivational interviewing (MI) techniques. The intervention targets HIV-positive African-American adults in inner-city Baltimore, Maryland who are suboptimally engaged in care and who endorse conspiracy beliefs about HIV or low readiness to begin ART.

In this project the investigators will conduct a small randomized controlled pilot trial to test the potential efficacy of PATCH in producing positive attitudinal changes, including a reduction in conspiracy beliefs and perceived barriers to ART and an increase in stated readiness to begin ART. The investigators will compare PATCH to an attentional control. Participants will be recruited from outpatient HIV clinics settings but will be individuals who are not taking ART. Assessments will be conducted at baseline, post-treatment (estimated 4-8 weeks post-baseline), and at 3-month post-baseline follow-up. The specific aims are: (1) Develop and refine a manual for a brief MI intervention to support ART decision-making and reduce the likelihood of ART refusal: (2) Evaluate the feasibility and acceptability of implementing the PATCH intervention in a small sample of individuals who are African-American, recommended for ART but who are not current taking it, and who experience multiple barriers to ART adherence; and (3) Conduct a small randomized controlled pilot to test the potential efficacy of the PATCH intervention in producing positive attitudinal changes, including a reduction in conspiracy beliefs and perceived barriers to ART and stated readiness to begin ART.

ELIGIBILITY:
Inclusion Criteria:

* Known to the recruitment site to be HIV-positive
* African-American or multiracial with African-American heritage.
* Able to speak and understand English.
* At least one of the following:

  1. Sub-optimally involved in HIV care (defined as no regular source of HIV primary care, clinically eligible for ART but not taking it, or received an offer of ART in the last year but not currently taking it.
  2. Non-adherent to ART (defined as being offered ART but not taking it or not appropriately adhering to it (as reflected by a score of 10 or less on screening questionnaire) at the time of enrollment.
  3. Conspiracy beliefs (defined as a score of 10 or more on screening questionnaire or states that would not be ready to take ART if recommended).

Exclusion Criteria:

* Known diagnosis of mental retardation or dementia.
* Active psychosis or suicidality evident in initial interview.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
positive attitudinal changes | baseline, week 6
  Positive attitudinal changes includes a reduction in conspiracy beliefs and perceived barriers to ART. Attitudes will be assessed via questionnaires completed at the baseline, post treatment, and follow-up assessments.
Stated readiness to begin ART | baseline, week 6
  Stated readiness to begin ART will be assessed via questionnaires and interviews completed at the post treatment assessment.

SECONDARY OUTCOMES:
Beginning ART | baseline, week 16
  Beginning ART will be assessed via questionnaires and interviews completed at the follow-up assessment, as well as by review of the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie E Bennett, Ph.D., Principal Investigator — University of Maryland, Baltimore; Seth Himelhoch, Md, MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States